CLINICAL TRIAL: NCT03809338
Title: Evaluation of Antral Follicle Count and Amh Values in Women Working at Night and Flight Attendants
Brief Title: Ovarian Functions in Flight Attendants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acibadem Fulya Hastanesi (Network)
Responsible Party: Sponsor
Other Study IDs: AcibademFulyaH
Record Dates: First submitted 2019-01-17; First posted 2019-01-18 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Ovarian Functions in Flight Attendants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 5 ml blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- flight attendant women: Assesment antral follicle count on day 3 5ml blood sample to be taken
  Interventions: Diagnostic Test: amh test
- day working women: Assesment antral follicle count on day 3 5ml blood sample to be taken
  Interventions: Diagnostic Test: amh test

INTERVENTIONS:
Diagnostic Test: amh test — Antral follicle count with ultrasound on the 3rd day of menstruation
  Other Names: Day 3 antral follicle with transvaginal ultrasonography

SUMMARY:
The aim of this study was to evaluate the effects of night sleep disorder and sleeplessness, excessive hours spent on flight and UV radiation exposure over ovarian function in flight attendant women.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effects of night sleep disorder and sleeplessness, excessive hours spent on flight and UV radiation exposure over ovarian function in flight attendant women.

On the third day of the menstrual period, evaluate the number of antral follicle count will be examined and the level of hormones showing the ovarian functions will be measured in the blood sample given by the participant.

ELIGIBILITY:
Inclusion Criteria:

* day working women , 25-35 years old
* night working women , 25-35 years old
* flight attendant women, 25-35 years old

Exclusion Criteria:

* those who cannot enter the groups above

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — evaluation ovarian functions of women
Study Population: 50 flight attendants and 50 control patients
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
level of amh | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem Fulya Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No